CLINICAL TRIAL: NCT06578962
Title: Evaluation of the Effects of Shampoo RV3438G in Recurrent Squamous States and Maintenance of the Effects
Brief Title: Efficacy of a Cosmetic Shampoo RV3438G in Reccurent Squamous States
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV3438G2020043
Record Dates: First submitted 2024-04-30; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Dermatitis, Seborrheic
Keywords: Dermatitis, Seborrheic; Scalp; Adults; Maintenance of effects
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab sampling of the scalp and cigarette paper sample on the target lesions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tested product RV3438G associated with gentle balancing shampoo
  Interventions: Other: Phase 1: short intensive treatment phase; Other: Phase 2 : Tested product RV3438G associated with gentle balancing shampoo
- Tested product RV3438G associated with neutral shampoo
  Interventions: Other: Phase 1: short intensive treatment phase; Other: Phase 2 : Tested product RV3438G associated with neutral shampoo
- Control group
  Interventions: Other: Phase 1: short intensive treatment phase; Other: Phase 2 : neutral shampoo

INTERVENTIONS:
Other: Phase 1: short intensive treatment phase — During the treatment phase (phase 1), all subjects of the study applied the tested product RV3438G, thrice a week, for 2 weeks.
Other: Phase 2 : Tested product RV3438G associated with gentle balancing shampoo — During maintenance phase (phase 2):
  the tested product RV3438G was applied once a week for 8 weeks the gentle balancing shampoo RD1089O was applied twice a week alternately with the RV3438G shampoo, for 8 weeks.
  Groups: Tested product RV3438G associated with gentle balancing shampoo
Other: Phase 2 : Tested product RV3438G associated with neutral shampoo — During maintenance phase (phase 2):
  the tested product RV3438G was applied once a week for 8 weeks the neutral shampoo RD0057H was applied twice a week alternately with the RV3438G shampoo, for 8 weeks.
  Groups: Tested product RV3438G associated with neutral shampoo
Other: Phase 2 : neutral shampoo — During maintenance phase (phase 2):
  the neutral shampoo RD0057H was applied thrice a week for 8 weeks.
  Groups: Control group

SUMMARY:
The aim of the study is to evaluate, with clinical, biological and biometrological assessment methods, the effectiveness of RV3438G shampoo, after 2 weeks of short intensive treatment phase and also the effects of a maintenance phase of 8 weeks in association with a neutral shampoo, or with a gentle balancing shampoo, compared to a neutral shampoo used single.

This is a bicentric, comparative (during the maintenance phase), randomized, controlled and open study, in parallel groups conducted in subjects having mild to moderate recurrent squamous states, for 10 weeks.

4 visits are planned. The maximum duration of the study is 74 days from inclusion visit to the End-of-study visit.

The study area is the whole scalp.

DETAILED DESCRIPTION:
4 visits are performed: Visit 1: Inclusion (Day1) : start of the short intensive treatment phase (phase 1) Visit 2: Intermediate visit (Day15 ± 3 days, Week 2) : end of the short treatment intensive phase and start of the maintenance phase (phase 2) Visit 3: Intermediate visit (Day 43 ± 3 days, Week 6) : middle of the maintenance phase Visit 4: End-of-study visit (Day 71 ± 3 days, Week 10) : end of the maintenance phase

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the population:

- Subject aged between 18 and 60 years included

Criteria related to the disease:

Subject having a squamous state of the scalp :

* clinically visible (Squire score ≥ 20),
* with an intensity of the squamous state superior or equal to 2 on a scale from 0 to 3 on at - least 1 of the 4 scalp areas
* recurrent (at least twice a year)
* associated to erythema and pruritus: erythema scoring superior or equal to 1 on a scale from 0 to 3 on at least 1 scalp area desquamating of the 4 scalp areas pruritus scoring assessed by the subject superior or equal to 3 on a numerical scale from 0 to 10 (mean pruritus felt on the last 3 days)

Exclusion Criteria:

Criteria related to the diseases / skin condition:

* Subject having frizzy hair
* Subject with an alopecia having caused hair loss on the upper part of the scalp (Norwood Hamilton stage> III, Ludwig ≥ I-4, alopecia aerata, alopecia totalis), Seborrheic dermatitis requiring medical treatment

Criteria related to treatments and/or products:

* Systemic treatment with nonsteroidal anti-inflammatory, corticosteroid, antibiotic, antihistamine taken during 5 consecutive days within the 2 weeks before the inclusion or planned during the study and liable to interfere with the study assessments
* Topical treatment or product applied on the scalp within 2 weeks before the inclusion or planned during the study that can be active on squamous states or that can limit the effectiveness of the study product: anti-inflammatory drugs, ketoconazole, anti-dandruff shampoo, anti-fungal, rinse with vinegar, essential oils ...
* Any scalp dyeing, bleaching, perm, smoothing / straightening performed within 2 weeks before inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be recruited from the panel of volunteers of the centre. The subjects corresponding to eligibility criteria may receive a phone call, a letter or an e-mail proposing to participate to the clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of the test product RV3438G during the maintenance phase by the global evolution of the squamous state assessed by the investigator | Assessed after 8 weeks of use, during the maintenance phase
  Dandruff score, from 0 to 80, calculated by the investigator with intensity (= severity, score from 1 to 5) x extent (= area, score from 0 to 4), for each quadrant of the scalp

SECONDARY OUTCOMES:
Efficacy of the test product RV3438G during the treatment phase by the global evolution of the squamous state assessed by the investigator | Assessed at baseline and after 2, 6 and 10 weeks of use
  Dandruff score, from 0 to 80, calculated by the investigator with intensity (= severity, score from 1 to 5) x extent (= area, score from 0 to 4), for each quadrant of the scalp
Efficacy of the test product RV3438G by the erythema evolution of the squamous state assessed by the investigator | assessed at baseline and after 2, 6 and 10 weeks of use
  assessed by the investigator on the scalp on a 4-point scale (from absent to severe)
Efficacy of the test product RV3438G by the pruritus evolution of the squamous state assessed by the subject | assessed at baseline and after 2, 6 and 10 weeks of use and weekly at home
  assessed by the subject on the scalp on a 10-point scale (from absent to maximal severity)
Efficacy of the test product RV3438G by the global evolution of the squamous state assessed by the investigator | assessed after 2, 6 and 10 weeks of use
  assessed by the investigator on the scalp on a 5-point scale (from worsening to complete resolution)
Efficacy of the test product RV3438G by the global evolution of the squamous state assessed by the subject | assessed weekly at home
  assessed by the subject on the scalp on a 5-point scale (from worsening to complete resolution)
Efficacy of the test product RV3438G by the evolution of the squamous state assessed by the subject | assessed at baseline and after 2, 6 and 10 weeks of use
  assessed by the subject on the scalp on a 4-point scale (from absent to severe)
Efficacy of the test product RV3438G by the evolution of the scalp discomfort assessed by the subject | assessed at baseline and weekly at home
  assessed by the subject on the scalp on a 4-point scale (from absent to severe)
Efficacy of the test product RV3438G by the analysis of skin microbiota diversity from scalp swab samples | assessed at baseline and after 2 and 10 weeks of use
  Microbiota diversity is analyzed by 16S and ITS1 sequencing.
Efficacy of the test product RV3438G by the analysis of skin microbiota composition from scalp swab samples | assessed at baseline and after 2, 6 and 10 weeks of use
  Microbiota composition is analyzed by ddPCR of some fungal and bacterial species
Efficacy of the test product RV3438G by the analysis of Inflammatory marker evolution from scalp swab samples | assessed at baseline and after 2 and 10 weeks of use
Efficacy of the test product RV3438G by the analysis of prurit marker evolution from scalp swab samples | assessed at baseline and after 2 and 10 weeks of use
Efficacy of the test product RV3438G by the analysis of cellular cohesion proteins evolution from scalp swab samples | assessed at baseline and after 2 and 10 weeks of use
Efficacy of the test product RV3438G by the Metabolomic analysis from scalp swab samples | assessed at baseline and after 2 and 10 weeks of use
Efficacy of the test product RV3438G by the analysis of molecular profiles of lipids from scalp cigarette paper sample | assessed at baseline and after 2, 6 and 10 weeks of use
  Assessed by FTIR analysis
Compliance of the subjects to the test product RV3438G | through study completion, 10 weeks
  The subject will report his/her compliance in a subject's diary
Tolerance of the test product RV3438G assessed by the investigator | assessed at baseline and after 2, 6 and 10 weeks of use
  Determined by the subject's spontaneous reporting, the investigator's non-leading questioning and his/her clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pascal REYGAGNE, Dr, Principal Investigator — Centre de santé SABOURAUD - Hôpital Saint Louis
Locations (1):
- Centre de Santé Sabouraud - Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maitre M, Baradat S, Froliger M, Turlier V, Simcic-Mori A, Gravier E, Genies C, Lauze C, Huyghe C, Noustens A, Alvarez-Georges S, Marinescu R, Reygagne P, Bessou-Touya S, Mengeaud V, Duplan H. Scalp Microbiome Dynamics Can Contribute to the Clinical Effect of a Novel Antiseborrheic Dermatitis Shampoo Containing Patented Antifungal Actives: A Randomized Controlled Study. Dermatol Ther (Heidelb). 2025 Aug;15(8):2077-2097. doi: 10.1007/s13555-025-01408-z. Epub 2025 Jun 11. PMID 40498389